CLINICAL TRIAL: NCT04329546
Title: How Immune Responses Shape Virological and Clinical Characteristics of COVID-19: a Prospective Cohort Study
Brief Title: Understanding COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Siegrist Claire-Anne, Professor of vaccinology, University Hospital, Geneva
Other Study IDs: 2020-00516
Record Dates: First submitted 2020-03-29; First posted 2020-04-01 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: SARS-CoV-2 Viral Kinetics and Host Immune Responses
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — naso- & oro-pharyngeal smears, sputum, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Cases are patients with COVID-19.
  Interventions: Other: NA (no intervention)
- Contacts: Contacts are household contacts of an index (case) patient.
  Interventions: Other: NA (no intervention)

INTERVENTIONS:
Other: NA (no intervention) — NA (no intervention)

SUMMARY:
This single-center prospective observational study will examine immune responses to to SARS-CoV-2 and how they correlate with its virological characteristics and clinical manifestations in infected patients. Household contacts will also be included so that early immune responses and viral kinetics can be captured. Patients and contacts will be followed for 8 and 2 weeks, respectively. The study will include a maximum of 250 participants.

DETAILED DESCRIPTION:
The primary aim of this single-center prospective observational study is to establish how immune responses to SARS-CoV-2 or to cross-reactive viruses correlate with the virological and clinical characteristics of SARS- CoV-2-infected patients and their exposed household contacts. Through iterative sampling, the viral kinetics of at least 50 infected patients will be evaluated in relation to symptom severity and innate and adaptive immune responses, while their household contacts will be observed for viral detection and immune responses. Patients and contacts will be followed for 8 and 2 weeks, respectively. The study will include a maximum of 250 participants.

ELIGIBILITY:
Inclusion Criteria:

The following persons may be included:

* A patient of any age meeting the European Centre for Disease Control and Prevention's confirmed case definition: "A person with laboratory confirmation of virus causing COVID-19, irrespective of clinical signs and symptoms" (and/or high suspicion/actively being treated as CoVID+ cases pending test confirmation)
* Household contacts (defined as those sleeping in the same apartment/house as an infected patient) of a patient with laboratory-confirmed COVID-19 (and/or high suspicion/actively being treated as CoVID+ cases pending test confirmation), whether symptomatic or not, and whether testing positive or not during a period of 14 days

Exclusion Criterion:

* Long-term incapacity leading to the inability to provide informed consent while not having a patient representative with the ability to provide informed consent

Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Adults and children of all ages either infected with, or presumed to be infected with SARS-CoV-2, and their household contacts.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Immunogenicity primary outcome: Geometric mean antibody concentration of total IgG antibodies to SARS-CoV-2 assessed by ELISA at 28 days | assessed at 28 days after diagnosis/presumed diagnosis
  Geometric mean antibody concentration of total IgG antibodies to SARS-CoV-2 assessed by ELISA at 28 days after diagnosis/suspected diagnosis
Virologic primary outcome: Peak viral load in the 56 days following diagnosis/suspected diagnosis | 56 days after diagnosis/presumed diagnosis
  Peak viral load in the 56 days following diagnosis/suspected diagnosis, quantified by real-time reverse-transcriptase polymerase chain reaction (RT-PCR) on nasopharyngeal swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Claire-Anne Siegrist, MD, Principal Investigator — Professor of vaccinology
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Fully anonymized data that are not already published may be shared on reasonable request from a qualified investigator, at the discretion of the Project Leader.